## Continue or Stop Applying Wet Cupping (Al-Hijamah) in Migraine Headache: A Non-Randomized Control Trial

Date:December 3<sup>rd</sup> 2017

## Statistical analysis

Analyses of the study data were made using SPSS vn 17.0 software. At the first stage of evaluation, descriptive statistics were applied and the age, gender, duration of pain and migraine type of the groups were stated as mean  $\pm$  standard deviation (SD) values. Conformity to normal distribution of the data was assessed with the Kolmogorov-Smirnov test. In groups showing normal distribution, the Student's t-test was used in the comparison of parametric data and the Chi-square test was used in the comparison of non-parametric data. In the comparisons of pre and post-treatment data within the groups, the Paired Samples t-test was used. A value of p<0.05 was accepted as statistically significant.